CLINICAL TRIAL: NCT06408818
Title: Online Parent Media Literacy Program to Promote Preadolescent Health
Brief Title: Study of an Online Program to Help Parents Talk With Their Tween Children About Health, Gender, Body-Image, and Relationships
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Innovation Research & Training (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TweenHealthStudy-R21-23-006-01; 5R21HD108440-02 (NIH)
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Results first posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-06

CONDITIONS: Parenting; Parent-Child Relations; Communication
Keywords: Preadolescent Health; Media Literacy; Parent-Child Communication; Gender Stereotypes; Body-Image; Puberty; Sexual Health; Relationship Health
MeSH Terms: conditions — Communication

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Program: Media Aware Parent -Tween (Experimental): Participants will have access to an intervention between pre-test and post-test assessments. The intervention, Media Aware Parent -Tween, is an online program for parents of tweens ages 9-12 designed to help parents have effective conversations with their child about body image, sexual development, gender stereotypes, romantic relationships, and media.
  Interventions: Behavioral: Media Aware Parent - Tween
- Active Control Resource (Active Comparator): Parents will have access to medically-accurate information about topics such as body image, sexual development, gender stereotypes, and romantic relationships.
  Interventions: Behavioral: Active Control Resource

INTERVENTIONS:
Behavioral: Media Aware Parent - Tween — Media Aware Parent - Tween, is an online program for parents of tweens ages 9-12 designed to help parents have effective conversations with their child about body image, sexual development, gender stereotypes, romantic relationships, and media.
  Arms: Intervention Program: Media Aware Parent -Tween
Behavioral: Active Control Resource — Parents will have access to medically-accurate information about topics such as body image, sexual development, gender stereotypes, and romantic relationships.
  Arms: Active Control Resource

SUMMARY:
The goal of this study is to learn if Media Aware Parent - Tween, an online program for parents of children ages 9-12, helps parents have effective conversations with their child about health and media.

DETAILED DESCRIPTION:
Parent-child pairs (N=300 pairs) will be recruited to participate in a randomized controlled trial. Parent consent and parent permission and youth assent will be sought. Participant pairs will be randomized into one of two study arms: intervention and active control. All participants will complete a web-based pre-test questionnaire. Youth and parents will then receive access to their randomly assigned resource. Approximately four weeks after completing the pre-test questionnaire, all participants will complete a web-based post-test questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* The adult must be the legal guardian of a child ages 9 to 12 years old.
* The parent must be able and willing to receive email and text communication as part of the study.
* The parent-child pair must have access to a smartphone with internet connection as the resource review will be completed online in a format that is best viewed on a smartphone.
* The parent-child pair must be fluent in English as the study materials are written in English.
* The parent must indicate that they will give the child participant privacy to complete the questionnaires.
* Both the adult and child must agree to participate.

Exclusion Criteria:

* Only one parent-child pair per family may participate in the study. If the parent has more than one child aged 9 to 12 that is willing to participate, the parent will be prompted to select the child participant based on the following: if the parent's last name begins with a letter from A to M, select the youngest eligible child willing to participate or if the parent's last name begins with a letter from N to Z, select the oldest eligible child willing to participate.
* In an effort to ensure diversity in parent gender and race/ethnicity, not all eligible pairs who are interested in participating will be enrolled in the study.

Min Age: 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 390 (Actual)
Dates: Start 2024-05-06 (Actual); Primary Completion 2025-03-24 (Actual); Study Completion 2025-03-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- innovation Research and Training, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Program: Media Aware Parent -Tween | Active Control Resource
Started (Total participants completed pretest (parent and child)) | 196 | 194
Parent Completed Pretest | 98 | 97
Child Completed Pretest | 98 | 97
Parent Completed Posttest | 91 | 88
Child Completed Posttest | 90 | 89
Completed (Total participants completed posttest (parent and child)) | 181 | 177
Not Completed | 15 | 17

BASELINE CHARACTERISTICS:
Population: Parents and children who were eligible and completed pretest. (Intervention included 98 parent-child pairs and control included 97 parent-child pairs)
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Program: Media Aware Parent -Tween | Active Control Resource | Total
Number analyzed (Participants) | 196 | 194 | 390
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: One parent from each condition was missing data on parent age.
  years
    Parents: number analyzed (Participants) | 97 | 96 | 193
    Parents | 40.79 (6.89) | 40.98 (6.72) | 40.89 (6.79)
    Children: number analyzed (Participants) | 98 | 97 | 195
    Children | 10.87 (1.01) | 10.55 (1.07) | 10.71 (1.05)
Sex/Gender, Customized [Number; unit: participants] — Population: Data for one child was missing in Intervention group.
  participants
    Parent Male: number analyzed (Participants) | 195 | 194 | 389
    Parent Male | 18 | 23 | 41
    Parent Female: number analyzed (Participants) | 195 | 194 | 389
    Parent Female | 80 | 74 | 154
    Parent Non-binary: number analyzed (Participants) | 195 | 194 | 389
    Parent Non-binary | 0 | 0 | 0
    Child Male: number analyzed (Participants) | 195 | 194 | 389
    Child Male | 43 | 40 | 83
    Child Female: number analyzed (Participants) | 195 | 194 | 389
    Child Female | 54 | 53 | 107
    Child Non-binary: number analyzed (Participants) | 195 | 194 | 389
    Child Non-binary | 0 | 4 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The overall sample size includes parents and children combined. The demographics were broken out by parent and child.
  Participants
    Parent: number analyzed (Participants) | 98 | 97 | 195
    Parent: Hispanic or Latino | 17 | 16 | 33
    Parent: Not Hispanic or Latino | 81 | 81 | 162
    Parent: Unknown or Not Reported | 0 | 0 | 0
    Child: number analyzed (Participants) | 98 | 97 | 195
    Child: Hispanic or Latino | 21 | 20 | 41
    Child: Not Hispanic or Latino | 77 | 77 | 154
    Child: Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The overall sample size includes parents and children combined. The demographics were broken out by parent and child.
  Participants
    Parents: number analyzed (Participants) | 98 | 97 | 195
    Parents: American Indian or Alaska Native | 3 | 1 | 4
    Parents: Asian | 5 | 10 | 15
    Parents: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Parents: Black or African American | 16 | 22 | 38
    Parents: White | 61 | 57 | 118
    Parents: More than one race | 3 | 1 | 4
    Parents: Unknown or Not Reported | 10 | 6 | 16
    Children: number analyzed (Participants) | 98 | 97 | 195
    Children: American Indian or Alaska Native | 2 | 1 | 3
    Children: Asian | 3 | 7 | 10
    Children: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Children: Black or African American | 18 | 20 | 38
    Children: White | 55 | 51 | 106
    Children: More than one race | 11 | 12 | 23
    Children: Unknown or Not Reported | 9 | 6 | 15
Region of Enrollment [Number; unit: participants]
  United States | 196 | 194 | 390

OUTCOME MEASURES:

1. Primary Outcome: Change From Pretest in Child Report of Frequency of Parent-child Communication
Description: Child will respond to questions about the frequency with which their parent has talked with them about 12 topics related to prepubescent health on a Likert-type scale [1 = Never; 2 = A little; 3 = A lot]. Reponses on items are averaged, and higher scores indicate a more favorable outcome.
Time Frame: Pretest (at baseline) and Posttest (about four weeks after pretest questionnaire completion)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention Program: Media Aware Parent -Tween | Active Control Resource
Number analyzed (Participants) | 98 | 97
score on a scale | 2.18 (0.05) | 2.20 (0.04)
Statistical Analysis 1: Comparison: Intervention Program: Media Aware Parent -Tween vs Active Control Resource; Test type: Equivalence — To examine intervention effects on primary outcomes at posttest, we used linear regression in intent-to-treat analyses. Posttest scores were regressed onto pretest scores, covariates, and the treatment effect; p = 0.69, Regression, Linear; Mean Difference (Final Values) = -0.02, Standard Error of Mean 0.06

2. Primary Outcome: Change From Pretest in Parent Report of Frequency of Parent-child Communication
Description: Parent will respond to questions about the frequency with which they have talked with their child about 12 topics related to prepubescent health on a Likert-type scale [1 = Never; 2 = A little; 3 = A lot]. Reponses on items are averaged, and higher scores indicate a more favorable outcome.
Time Frame: Pretest (at baseline) and Posttest (about four weeks after pretest questionnaire completion)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention Program: Media Aware Parent -Tween | Active Control Resource
Number analyzed (Participants) | 98 | 97
score on a scale | 2.42 (0.03) | 2.37 (0.04)
Statistical Analysis 1: Comparison: Intervention Program: Media Aware Parent -Tween vs Active Control Resource; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.33, Regression, Linear; Mean Difference (Final Values) = 0.05, Standard Error of Mean 0.05

3. Primary Outcome: Change From Pretest in Child Report of General Parent-child Communication Quality
Description: Child will indicate the extent to which they agree with nine statements about communication with their parent on a Likert-type scale [1 = Strongly disagree, 2 = Disagree, 3 = Agree, 4 = Strongly agree]. Reponses on items are averaged, and higher scores indicate a more favorable outcome.
Time Frame: Pretest (at baseline) and Posttest (about four weeks after pretest questionnaire completion)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention Program: Media Aware Parent -Tween | Active Control Resource
Number analyzed (Participants) | 98 | 97
score on a scale | 2.97 (0.05) | 3.02 (0.05)
Statistical Analysis 1: Comparison: Intervention Program: Media Aware Parent -Tween vs Active Control Resource; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.46, Regression, Linear; Mean Difference (Final Values) = -0.05, Standard Error of Mean 0.07

4. Primary Outcome: Change From Pretest in Parent Report of General Parent-child Communication Quality
Description: Parent will indicate the extent to which they agree with nine statements about communication with their child on a Likert-type scale [1 = Strongly disagree, 2 = Disagree, 3 = Agree, 4 = Strongly agree]. Reponses on items are averaged, and higher scores indicate a more favorable outcome.
Time Frame: Pretest (at baseline) and Posttest (about four weeks after pretest questionnaire completion)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention Program: Media Aware Parent -Tween | Active Control Resource
Number analyzed (Participants) | 98 | 97
score on a scale | 3.08 (0.04) | 3.12 (0.04)
Statistical Analysis 1: Comparison: Intervention Program: Media Aware Parent -Tween vs Active Control Resource; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.46, Regression, Linear; Mean Difference (Final Values) = -0.04, Standard Error of Mean 0.06

5. Primary Outcome: Change From Pretest in Child Report of Active Parental Media Mediation
Description: Child's perception of parent's use of active media mediation will be assessed using two items (e.g., "How often does your parent tell you what they see in media is different than real life?"). Participants will rate items on a 5-point Likert scale [1 = never; 2 = almost never; 3 = sometimes; 4 = often; 5 = very often]. Reponses on items are averaged, and higher scores indicate a more favorable outcome.
Time Frame: Pretest (at baseline) and Posttest (about four weeks after pretest questionnaire completion)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention Program: Media Aware Parent -Tween | Active Control Resource
Number analyzed (Participants) | 98 | 97
score on a scale | 3.46 (0.12) | 3.69 (0.12)
Statistical Analysis 1: Comparison: Intervention Program: Media Aware Parent -Tween vs Active Control Resource; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.20, Regression, Linear; Mean Difference (Final Values) = -0.22, Standard Error of Mean 0.17

6. Primary Outcome: Change From Pretest in Parent Report of Active Parental Media Mediation
Description: Parents' use of active media mediation will be assessed using two items (e.g., "How often do you tell your child what they see in media is different than real life?"). Participants will rate items on a 5-point Likert scale [1 = never; 2 = almost never; 3 = sometimes; 4 = often; 5 = very often]. Reponses on items are averaged, and higher scores indicate a more favorable outcome.
Time Frame: Pretest (at baseline) and Posttest (about four weeks after pretest questionnaire completion)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention Program: Media Aware Parent -Tween | Active Control Resource
Number analyzed (Participants) | 98 | 97
score on a scale | 4.17 (0.07) | 4.04 (0.08)
Statistical Analysis 1: Comparison: Intervention Program: Media Aware Parent -Tween vs Active Control Resource; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.22, Regression, Linear; Mean Difference (Final Values) = 0.13, Standard Error of Mean 0.11

7. Primary Outcome: Change From Pretest in Child Report of Parental Restrictive Media Mediation
Description: Child's perception of parent's use of restrictive media mediation will be assessed using one item (e.g., "How often does your parent limit the amount of your screen time (watching shows, going online, playing video games, or using social media)?"). Participants will rate items on a 5-point Likert scale [1 = never; 2 = almost never; 3 = sometimes; 4 = often; 5 = very often]. Higher scores indicate a more favorable outcome.
Time Frame: Pretest (at baseline) and Posttest (about four weeks after pretest questionnaire completion)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention Program: Media Aware Parent -Tween | Active Control Resource
Number analyzed (Participants) | 98 | 97
score on a scale | 3.70 (0.13) | 3.57 (0.13)
Statistical Analysis 1: Comparison: Intervention Program: Media Aware Parent -Tween vs Active Control Resource; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.48, Regression, Linear; Mean Difference (Final Values) = 0.13, Standard Error of Mean 0.19

8. Primary Outcome: Change From Pretest in Parent Report of Parental Restrictive Media Mediation
Description: Parent's use of restrictive media mediation will be assessed using one item (e.g., "How often do you limit the amount of your child's screen time (watching shows, going online, playing video games, or using social media)?"). Participants will rate items on a 5-point Likert scale [1 = never; 2 = almost never; 3 = sometimes; 4 = often; 5 = very often].
  Higher scores indicate a more favorable outcome.
Time Frame: Pretest (at baseline) and Posttest (about four weeks after pretest questionnaire completion)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention Program: Media Aware Parent -Tween | Active Control Resource
Number analyzed (Participants) | 98 | 97
score on a scale | 3.88 (0.11) | 3.81 (0.11)
Statistical Analysis 1: Comparison: Intervention Program: Media Aware Parent -Tween vs Active Control Resource; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.69, Regression, Linear; Mean Difference (Final Values) = 0.06, Standard Error of Mean 0.16

9. Primary Outcome: Change From Pretest in Child Report of Awareness of Family Media Rules
Description: Child will indicate on one item whether their family has rules about media use. Response options are "yes (1)," "no (0)," and "unsure (2)". Yes (1) indicates a more favorable outcome.
Time Frame: Posttest (about four weeks after pretest questionnaire completion)
Population: This analysis was conducted using multiple imputed data. Therefore, the percentage values will not yield a whole participant because results are pooled between 50 imputations.
Measure: Number; unit: percentage of participants with "1"
Arm/Group | Intervention Program: Media Aware Parent -Tween | Active Control Resource
Number analyzed (Participants) | 98 | 97
percentage of participants with "1" | 81.96 | 90.72
Statistical Analysis 1: Comparison: Intervention Program: Media Aware Parent -Tween vs Active Control Resource; Test type: Equivalence — To examine intervention effects on primary outcomes at posttest, we used logistic regression in intent-to-treat analyses. Posttest scores were regressed onto pretest scores, covariates, and the treatment effect; p = 0.22, Regression, Logistic; Mean Difference (Final Values) = -0.78, Standard Error of Mean 0.63

10. Primary Outcome: Change From Pretest in Parent Report of Awareness of Family Media Rules
Description: Parent will indicate on one item whether their family has rules about media use. Response options are "yes (1)," "no (0)," and "unsure (2)". Yes (1) indicates a more favorable outcome.
Time Frame: Posttest (about four weeks after pretest questionnaire completion)
Population: as for outcome 9
Measure: Number; unit: percentage of participants w/ "1"
Arm/Group | Intervention Program: Media Aware Parent -Tween | Active Control Resource
Number analyzed (Participants) | 98 | 97
percentage of participants w/ "1" | 89.88 | 92.89
Statistical Analysis 1: Comparison: Intervention Program: Media Aware Parent -Tween vs Active Control Resource; Test type: Equivalence — [test comment as in outcome 9, analysis 1]; p = 0.57, Regression, Logistic; Slope = -0.45, Standard Error of Mean 0.79

11. Primary Outcome: Change From Pretest in Child Report of Acceptance of Gender Stereotypical Roles
Description: Child will respond to the 7 items to indicate their agreement with statements about gender using a 5-point Likert scale (1 = "disagree a lot" to 5 = "agree a lot"). Reponses on items are averaged, and higher scores indicate a less favorable outcome.
Time Frame: Pretest (at baseline) and Posttest (about four weeks after pretest questionnaire completion)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention Program: Media Aware Parent -Tween | Active Control Resource
Number analyzed (Participants) | 98 | 97
score on a scale | 1.86 (0.07) | 1.77 (0.07)
Statistical Analysis 1: Comparison: Intervention Program: Media Aware Parent -Tween vs Active Control Resource; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.42, Regression, Linear; Mean Difference (Final Values) = 0.08, Standard Error of Mean 0.10

12. Primary Outcome: Change From Pretest in Child Report of Attitudes Toward Puberty
Description: Child will respond to one item (i.e., "I like the fact that I am becoming a woman/man") on a 4-point scale from 1 = disagree a lot to 4 = Agree a lot to assess participants' attitudes towards puberty. Higher scores indicate a more favorable outcome.
Time Frame: Pretest (at baseline) and Posttest (about four weeks after pretest questionnaire completion)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention Program: Media Aware Parent -Tween | Active Control Resource
Number analyzed (Participants) | 98 | 97
score on a scale | 2.97 (0.09) | 3.07 (0.09)
Statistical Analysis 1: Comparison: Intervention Program: Media Aware Parent -Tween vs Active Control Resource; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.45, Regression, Linear; Mean Difference (Final Values) = -0.10, Standard Error of Mean 0.13

13. Primary Outcome: Change From Pretest in Child Report of Body-esteem
Description: Child will respond to four statements about how they feel about their body (e.g., I'm proud of my body) on a 5-point scale [1 = Never; 2 = Seldom; 3 = Sometimes; 4 = Often; 5 =Always]. Reponses on items are averaged, and higher scores indicate a more favorable outcome.
Time Frame: Pretest (at baseline) and Posttest (about four weeks after pretest questionnaire completion)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention Program: Media Aware Parent -Tween | Active Control Resource
Number analyzed (Participants) | 98 | 97
score on a scale | 3.32 (0.09) | 3.42 (0.08)
Statistical Analysis 1: Comparison: Intervention Program: Media Aware Parent -Tween vs Active Control Resource; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.39, Regression, Linear; Mean Difference (Final Values) = -0.10, Standard Error of Mean 0.12

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from pretest to posttest completion: approximately 4 weeks.
Description: Participants were grouped as dyads for the purposes of recruitment and analyses. Therefore, parent and child were grouped when reporting adverse events. Notably, there were no adverse events to report in any dyads, including among both parents and children.
Arm/Group | Intervention Program: Media Aware Parent -Tween | Active Control Resource
All-Cause Mortality (participants affected / at risk) | 0/196 | 0/194
Serious Adverse Events (participants affected / at risk) | 0/196 | 0/194
Other Adverse Events (participants affected / at risk) | 0/196 | 0/194

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-22): https://cdn.clinicaltrials.gov/large-docs/18/NCT06408818/Prot_SAP_000.pdf